CLINICAL TRIAL: NCT05301647
Title: Mometasone Furoate Nasal Spray in Italian Children With Seasonal Allergic Rhinitis: a Comprehensive Assessment
Brief Title: Mometasone Furoate Nasal Spray in Italian Children
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Prof. Michele Miraglia del Giudice, Associate professor, University of Campania Luigi Vanvitelli
Other Study IDs: VANVCIT1
Record Dates: First submitted 2022-03-01; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Rhinitis, Allergic; Nasal Allergy; Allergy Pollen; Nasal, Cytology; Mometasone Allergy; Quality of Life; Child, Only
Keywords: seasonal allergic rhinitis; mometasone furoate nasal spray; nasal cytology; type 2 inflammation; symptoms; quality of life
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active Group
  Interventions: Diagnostic Test: Nasal cytology; Other: The validated Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ); Other: Total symptom score (TSS); Other: Visual analogic scale (VAS)
- Control Group
  Interventions: Diagnostic Test: Nasal cytology; Other: The validated Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ); Other: Total symptom score (TSS); Other: Visual analogic scale (VAS)

INTERVENTIONS:
Diagnostic Test: Nasal cytology — The cytological technique involves the following moments: sampling, processing, which includes fixation, staining and microscopic observation. Cytological sampling consists in the collection of superficial cells of the nasal mucosa with the help of a sterile swab or a small curette (scraping) in disposable plastic material (Rhino-probe).
Other: The validated Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) — The validated Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) consists of 23 questions in 5 domains (nasal symptoms, ocular symptoms, practical issues, limitation of activities, other symptoms) that are answered on a 7-point scale (0-6), where 0 represents the absence of problems and 6 the greatest symptom distress. Children will complete the questionnaire together with a parent at baseline and during the study. A Total Score was calculated as the mean of the 5 domains.
Other: Total symptom score (TSS) — Total symptom score was the sum of 3 domains: i) nasal symptoms (TNSS) included itching, sneezing, rhinorrhea, nasal congestion; ii) ocular symptoms (TOSS): itching, hyperemia of the conjunctiva, tearing; and iii) throat symptoms (TTSS): itching, coughing. With the help of their parents, patients scored symptoms severity on a 4-point scale: 0 = absent or irrelevant, 1 = mild, 2 = moderate, 3 = severe. Total symptom score was assessed at 12 hours (TTS 12h) and two weeks (TTS 2W) before the visits. TSS represents the doctor's point of view of symptom severity
Other: Visual analogic scale (VAS) — A visual analogic scale (VAS) measured the parental perception of symptom severity (0=no symptom; 10=very severe symptoms).

SUMMARY:
Objective Seasonal allergic rhinitis (SAR) is a common disease in childhood and characterized by type 2 inflammation, bothersome symptoms, and impaired quality of life (QoL). Intranasal corticosteroids are effective medications in managing SAR patients. In addition, mometasone furoate nasal spray (MFNS) is a well-known therapeutic option. However, the literature provided no data about its effects in European children with SAR. Thus this study addressed this unmet need.

DETAILED DESCRIPTION:
Objective Seasonal allergic rhinitis (SAR) is a common disease in childhood and characterized by type 2 inflammation, bothersome symptoms, and impaired quality of life (QoL). Intranasal corticosteroids are effective medications in managing SAR patients. In addition, mometasone furoate nasal spray (MFNS) is a well-known therapeutic option. However, the literature provided no data about its effects in European children with SAR. Thus this study addressed this unmet need.

Methods MFNS was compared to isotonic saline. Both treatments were prescribed one spray per nostril, twice a day, per 3 weeks. Nasal cytology, total symptom score (TSS), visual analogic scale concerning the parental perception of symptom severity, and the Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) were assessed at baseline, after 7 and 21 days, and one month after discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were: age range 4-12 years, SAR diagnosis, Total Symptoms Score (TSS) ≥ 6, and written informed consent of both parents or legal guardians.

Exclusion Criteria:

* Exclusion criteria were: perennial AR, rhinitis due to other causes, concomitant acute or chronic rhinosinusitis, nasal polyps, asthma comorbidity, current use of topical or systemic corticosteroids, antihistamines, antileukotrienes, inadequate washout of them, nasal anatomic defect, respiratory infections in the last two weeks, participation in other clinical studies in the previous month, documented hypersensitivity to the study product or its excipients, and trip planned outside of the study area.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Globally, 80 children were enrolled, but 76 (40 males and 36 females, mean age 11.4 + 3.3 years) completed the study. Children were randomly (ratio 1:1) subdivided into two groups: the active group treated with MFNS (Mometasone group) and the control group treated with isotonic saline.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Change in eosinophils, mast cells and neutrophil infiltrate by nasal cytology after the treatment | 2019-2021
  The primary endpoint of this study was the change in eosinophilic mast cells and neutrophil infiltrate, assessed by nasal cytology

SECONDARY OUTCOMES:
Assesment of symptoms during the study | 2019-2021
  The secondary objective was the nasal symptom severity during the study assessed by total symptom score (TSS)
Assesment of quality of life changes during the study | 2019-2021
  The secondary objective was the changes of quality of life during the study assessed by the validated Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Second University, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wise SK, Lin SY, Toskala E, Orlandi RR, Akdis CA, Alt JA, Azar A, Baroody FM, Bachert C, Canonica GW, Chacko T, Cingi C, Ciprandi G, Corey J, Cox LS, Creticos PS, Custovic A, Damask C, DeConde A, DelGaudio JM, Ebert CS, Eloy JA, Flanagan CE, Fokkens WJ, Franzese C, Gosepath J, Halderman A, Hamilton RG, Hoffman HJ, Hohlfeld JM, Houser SM, Hwang PH, Incorvaia C, Jarvis D, Khalid AN, Kilpelainen M, Kingdom TT, Krouse H, Larenas-Linnemann D, Laury AM, Lee SE, Levy JM, Luong AU, Marple BF, McCoul ED, McMains KC, Melen E, Mims JW, Moscato G, Mullol J, Nelson HS, Patadia M, Pawankar R, Pfaar O, Platt MP, Reisacher W, Rondon C, Rudmik L, Ryan M, Sastre J, Schlosser RJ, Settipane RA, Sharma HP, Sheikh A, Smith TL, Tantilipikorn P, Tversky JR, Veling MC, Wang Y, Westman M, Wickman M, Zacharek M. International Consensus Statement on Allergy and Rhinology: Allergic Rhinitis. Int Forum Allergy Rhinol. 2018 Feb;8(2):108-352. doi: 10.1002/alr.22073. PMID 29438602
- [Result] Wen T, Rothenberg ME. Cell-by-cell deciphering of T cells in allergic inflammation. J Allergy Clin Immunol. 2019 Nov;144(5):1143-1148. doi: 10.1016/j.jaci.2019.10.001. PMID 31703761
- [Result] Han X, Krempski JW, Nadeau K. Advances and novel developments in mechanisms of allergic inflammation. Allergy. 2020 Dec;75(12):3100-3111. doi: 10.1111/all.14632. Epub 2020 Nov 4. PMID 33068299
- [Result] Ciprandi G, Klersy C, Cirillo I, Marseglia GL. Quality of life in allergic rhinitis: relationship with clinical, immunological, and functional aspects. Clin Exp Allergy. 2007 Oct;37(10):1528-35. doi: 10.1111/j.1365-2222.2007.02809.x. PMID 17883732
- [Result] Ciprandi G, Cirillo I, Vizzaccaro A, Milanese M, Tosca MA. Nasal obstruction in patients with seasonal allergic rhinitis: relationships between allergic inflammation and nasal airflow. Int Arch Allergy Immunol. 2004 May;134(1):34-40. doi: 10.1159/000077531. Epub 2004 Mar 25. PMID 15051938
- [Result] Cirillo I, Marseglia G, Klersy C, Ciprandi G. Allergic patients have more numerous and prolonged respiratory infections than nonallergic subjects. Allergy. 2007 Sep;62(9):1087-90. doi: 10.1111/j.1398-9995.2007.01401.x. Epub 2007 Jun 18. PMID 17578494
- [Result] Juel-Berg N, Darling P, Bolvig J, Foss-Skiftesvik MH, Halken S, Winther L, Hansen KS, Askjaer N, Heegaard S, Madsen AR, Opstrup MS. Intranasal corticosteroids compared with oral antihistamines in allergic rhinitis: A systematic review and meta-analysis. Am J Rhinol Allergy. 2017 Jan 9;31(1):19-28. doi: 10.2500/ajra.2016.30.4397. PMID 28234147
- [Result] Baldwin CM, Scott LJ. Mometasone furoate: a review of its intranasal use in allergic rhinitis. Drugs. 2008;68(12):1723-39. doi: 10.2165/00003495-200868120-00009. PMID 18681494
- [Result] Ciprandi G, Varricchio A. The relevance of the Mometasone furoate nasal spray in clinical practice. J Biol Regul Homeost Agents. 2018 Jul-Aug;32(4):1051-1054. PMID 30043593
- [Result] Meltzer EO, Baena-Cagnani CE, Gates D, Teper A. Relieving nasal congestion in children with seasonal and perennial allergic rhinitis: efficacy and safety studies of mometasone furoate nasal spray. World Allergy Organ J. 2013 Mar 4;6(1):5. doi: 10.1186/1939-4551-6-5. PMID 23663488
- [Result] Meltzer EO, Shekar T, Teper AA. Mometasone furoate nasal spray for moderate-to-severe nasal congestion in subjects with seasonal allergic rhinitis. Allergy Asthma Proc. 2011 Mar-Apr;32(2):159-67. doi: 10.2500/aap.2011.32.3424. PMID 21439168
- [Result] Ciprandi G, Tosca MA, Passalacqua G, Canonica GW. Intranasal mometasone furoate reduces late-phase inflammation after allergen challenge. Ann Allergy Asthma Immunol. 2001 Apr;86(4):433-8. doi: 10.1016/S1081-1206(10)62491-X. PMID 11345288
- [Result] Hoyte FCL, Nelson HS. Recent advances in allergic rhinitis. F1000Res. 2018 Aug 23;7:F1000 Faculty Rev-1333. doi: 10.12688/f1000research.15367.1. eCollection 2018. PMID 30210782
- [Result] Karatzas K, Katsifarakis N, Riga M, Werchan B, Werchan M, Berger U, Pfaar O, Bergmann KC. New European Academy of Allergy and Clinical Immunology definition on pollen season mirrors symptom load for grass and birch pollen-induced allergic rhinitis. Allergy. 2018 Sep;73(9):1851-1859. doi: 10.1111/all.13487. Epub 2018 Jun 17. PMID 29791010
- [Result] Gelardi M, Fiorella ML, Russo C, Fiorella R, Ciprandi G. Role of nasal cytology. Int J Immunopathol Pharmacol. 2010 Jan-Mar;23(1 Suppl):45-9. PMID 20152080
- [Result] Juniper EF, Guyatt GH, Feeny DH, Ferrie PJ, Griffith LE, Townsend M. Measuring quality of life in children with asthma. Qual Life Res. 1996 Feb;5(1):35-46. doi: 10.1007/BF00435967. PMID 8901365
- [Result] Benazzo M, Leonardi S, Corsico A, Licari A, Miraglia Del Giudice M, Peroni D, Salpietro C, Marseglia GL, Ciprandi G. Cetirizine modifies quality of life and symptoms in children with seasonal allergic rhinitis: a pilot study. Acta Biomed. 2020 Jun 17;92(1):e2021003. doi: 10.23750/abm.v92i1.9948. PMID 33682837
- [Result] Madison S, Brown EA, Franklin R, Wickersham EA, McCarthy LH. Clinical Question: Nasal saline or intranasal corticosteroids to treat allergic rhinitis in children. J Okla State Med Assoc. 2016 Apr-May;109(4-5):152-3. PMID 27328556

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT05301647/Prot_SAP_000.pdf